CLINICAL TRIAL: NCT01016613
Title: Clinical Phenotyping Resource and Biobank Core of the Michigan O'Brien Renal Center
Acronym: C-PROBE
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: St. John Health System, Michigan (Other); Temple University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Markus Bitzer, Professor of Medicine, University of Michigan
Other Study IDs: P30DK081943 (NIH); P30DK081943 (NIH)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Glomerulopathy
Keywords: chronic kidney disease; glomerulonephritis; proteinuria; nephrotic syndrome; nephropathy; biobank
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glomerulonephritis; Proteinuria; Nephrotic Syndrome; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood and renal tissue, if available
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Kidney Disease Cohort: chronic kidney disease patients with any type of kidney disease
- Matched Control Group: Healthy controls
- Trios: First degree relatives of pediatric chronic kidney disease cohort members

SUMMARY:
Chronic kidney disease (CKD) affects approximately 26 million Americans and disproportionately manifests in specific race and ethnic groups. Patients burdened with CKD have significant morbidity and reduced life expectancy. In addition to excessive suffering and lost productivity, the cost of managing this epidemic has reached $40 billion annually. The recognition that CKD is a major public health problem is reflected in the fourteen objectives outlined in Healthy People 2020 to begin to address the disease burden. Advancement in approaches to halt CKD progression has been slow despite growing global awareness of disease burden.

This O'Brien Kidney Research Core will create opportunities for novel insights through characterization of tissue profiles that will define new disease markers and molecular pathways and will be available to all kidney investigators on the www. It will thereby fundamentally alter the starting point for research into prevention of progression of these kidney diseases. C-PROBE is an essential element of the center grant and presents a biomedical resource core consisting of: (1) clinical phenotyping (that is, systematic identification of observable physical and biomedical characteristics) of kidney disease patients including the accurate measurement of kidney function; and (2) a specimen BioBank which will store blood, urine and kidney tissue samples. A key component of C-PROBE is therefore that it contains a proven mechanism to collect samples from high risk groups including minorities, at the institutions of University of Michigan Health System, St. John Hospital, Wayne State University in Michigan, John H. Stroger Hospital in Illinois, Temple University Health System in Pennsylvania, and Levine Children's Hospital in North Carolina. This mechanism will feed the other Cores and provide biomedical investigators with approved projects the access to a dynamic pool of well characterized high risk kidney disease patients and their biological specimens to conduct high caliber translational research.

ELIGIBILITY:
Inclusion Criteria:

* persons of any age who have chronic kidney disease (abnormally high protein in urine or reduced kidney function determined by blood tests)
* a small number of people without chronic kidney disease

Exclusion Criteria:

* people on hemodialysis or peritoneal dialysis
* people who have had a kidney transplant
* people unable or unwilling to provide consent
* women who are pregnant or nursing
* adults who have polycystic kidney disease
* institutionalized persons
* people currently participating in a blinded interventional clinical trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nephrology clinic patients and community members
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Subramanium Pennathur, MBBS, Principal Investigator — University of Michigan; Crystal A Gadegbeku, MD, Study Director — The Cleveland Clinic; Matthias Kretzler, MD, Study Director — University of Michigan; Markus Bitzer, MD, Study Director — University of Michigan
Locations (5):
- United States (5):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - St. John's Health System, Detroit, Michigan
  - Levine Children's Hospital, Charlotte, North Carolina
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No